CLINICAL TRIAL: NCT03942848
Title: Assessment of Intrathecal Ziconotide Antalgic Efficacy for Severe Refractory Neuropathic Pain Due to Spinal Cord Lesions.
Brief Title: Intrathecal Ziconotide Antalgic Efficacy for Severe Refractory Neuropathic
Acronym: SPIDOL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL18_0034
Record Dates: First submitted 2018-05-18; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Severe Refractory Neuropathic Pain; Spinal Cord Lesions
Keywords: Spinal cord lesion; intrathecal infusion; refractory neuropathic pain; ziconotide
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrathecal Ziconotide followed by placebo (Experimental): Each of the 44 patients will receive alternatively treatment or placebo, for 6 months. The treatment for each period will be randomly assigned. A washout period of 15 days will be applied between the two periods of infusion.
  Interventions: Drug: zicotinide followed by placebo; Drug: Placebo followed by zicotinide
- intrathecal Ziconotide preceded by placebo (Placebo Comparator): Each of the 44 patients will receive alternatively treatment or placebo, for 6 months. The treatment for each period will be randomly assigned. A washout period of 15 days will be applied between the two periods of infusion.
  Interventions: Drug: zicotinide followed by placebo; Drug: Placebo followed by zicotinide

INTERVENTIONS:
Drug: zicotinide followed by placebo — The experimental treatment period consists of Ziconotide solution that will be prepared by each local pharmacy team, in 5 or 10 milliliter (ml) vials with constant concentration of 10micrograms/mL
Drug: Placebo followed by zicotinide — The placebo treatment period consists in standard saline solution (preservative-free sodium chloride 9 milligram/milliliter (mg/ml) (0.9%) solution) which will be presented exactly in vials as presented for the treatment (volume, color, shape et size of the vial). Treating physicians will not be aware of the actual contents of the pump and will increase the volume of injected placebo as a treatment solution (as Ziconotide 10 micrograms/milliliter (μg/ml). The magnitude of increase is the decision of the treating physician (as long as it remains with the recommended limits by the Hospital Anxiety and Depression Scale (HAS) but most likely augmentations will be at maximum 1 microgram per month and maximum achieved doses allowed in SPIDOL study is 20 micrograms/day (in literature approximately 75% of patients who respond satisfactorily to treatment required a dose of ≤ 9.6 micrograms/day

SUMMARY:
Spinal cord injury (SCI) has an average prevalence of 50 per 100.000 in general population (30.000 patients with SCI in France) with estimates of the overall prevalence for severe neuropathic pain ranges from 30 to 51% (up to 10.000 patients in France).

Patients with such spinal lesions may develop neuropathic pain called sublesional pain as perceived in an area below the level of injury. A second type of pain is at level of injury, i.e. perceived in a segmental pattern within the dermatome corresponding the spinal cord and nerve roots. These two types of pain are very harmful and are notoriously difficult to treat probably because of complex pathogenic mechanisms due to abnormal functioning of deafferented spinal and supraspinal nociceptive neurons.

Opioids, whatever be the route of administration, had demonstrated their inefficacy for these patients as well as several surgical techniques. So, chronic pain in relation with spinal lesion can be defined as real refractory pain.

Synaptic release of neurotransmitters is dependent on calcium intake trough voltage dependent channels. Type 2.1 or N-Type channels are specific for nociceptive system and can be blocked by a peptic neurotoxin: Ziconotide. Blocking these specific calcium channels neuromodulates nociception. Intrathecal use of Ziconotide, bringing the active molecule close to its receptors, has a proven clinical impact for a wide variety of pain (4). The intrathecal Ziconotide (ITZ) infusion using an implanted pump is validated for treatment of pain refractory to systemic analgesics (HAS, avis du 14-27 mai 2008). Meanwhile, no data are available in literature on positive effects of ITZ on specific spinal neuropathic pain.

A pilot study was performed by the coordinator team using ITZ on 12 patients with spinal pain: 8 patients had > 40% decrease of pain on numeric scale, 6 patients beneficiated from implanted pump allowing chronic ITZ treatment inducing 60% numeric scale decrease in average with 1 year follow-up.

Therefore intrathecal Ziconotide could be an excellent candidate for the treatment of spinal pain where the pain generators may be difficult to target by other available treatments.

This study is the first to assess ITZ (as IT antalgic monotherapy) versus placebo with a randomized controlled study with long follow-up. Trials have already been performed but not specially targeted spinal pain, and did not exceed three weeks follow-up.

Long term effects of Ziconotide on memory, cognition and mood have not been evaluated. In fact even though short term adverse effects on higher level functions have been described they have not been assessed in a placebo controlled situation.

Moreover, treating (successfully or not) patients with spinal pain could bring valuable insights both into the mechanisms of pain production in SCI patients and in the mechanisms of Ziconotide action: a positive result on pain below the injury level would imply action on the second or third order synapses of the nociceptive pathways. Similarly an effect at the level of pain, in absence of an effect below the level pain would argue discussion against such action. The impact of ITZ on the different clinical components of pain experienced by the patients, could also give some data on neuromodulation mechanism induced by the therapy.

ELIGIBILITY:
Inclusion Criteria:

* • Patient > 18 year old

  * Patients with stabilized spinal cord lesion
  * Patients with refractory neuropathic pain with "Douleur Neuropathique" (DN4) score >4 at selection and failure at least of 2 classes of antineuropathic pain drugs alone or in association
  * Experiences pain > 5/10 on numeric scale
  * Patients with a positive trial test to Ziconotide either by lumbar puncture or by continuous infusion above the lesioned level via an implanted catheter
  * Evaluation performed both by a multidisciplinary team in a pain center and a rehabilitation center
  * Patients eligible to surgical implantation of a subcutaneous pump
  * Signed informed consent
  * Patients benefiting from a social insurance system or a similar system

Exclusion Criteria:

* • Life expectancy < 5 years

  * Suffering from other neuropathic pain or chronic pain due to cancer
  * Being treated with spinal cord stimulation, nerve stimulation, intrathecal analgesic delivery system with analgesic drug (except Baclofen) until the last 6 months
  * Implant ITZ surgery contraindication (MRI or anesthesia contraindication, coagulation disorder, Immunodepression, current infection, critical respiratory and/or heart illness)
  * Unable to operate the ITZ equipment or comply with study requirements
  * Suspicion of substance abuse
  * Current or planned pregnancy
  * Patients with urinary tract disorder or urinary retention
  * Patient under or planning to go under electromagnetic transcranial stimulation or planning to
  * Patient unable to understand the purpose of the trial or refusing to follow treatment and post-treatment instructions
  * Patients with history of psychiatric disorder or hallucination
  * Participation to another trial that would interfere with this trial
  * Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Change in pain between both treatment arms assessed by the Visual Analogic Scale (VAS) | 12 months
  The primary endpoint is the comparison, for each patient, of the mean pain intensity, within the last two week before the end of treatment, between two conditions: under Intrathecal Ziconotide (ITZ) and intrathecal (IT) placebo, using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of pain and 10 being the highest level of pain.The final endpoint will be measured after 6 months of treatment and 6 months of placebo (or vice versa according to the random assignation of first treatment in this cross over design study), that is to say after a total of 12 months of treatment.

SECONDARY OUTCOMES:
Evaluation of Long term analgesic effect of intrathecal Ziconotide assessed by the Visual Analogic Scale (VAS) | 12 months
  Continuous evaluation of pain intensity will be assessed using a visual analogic scale during the 12 months of treatment. Pain intensity will be measured using visual analogic scale (VAS). This VAS is a graduated line from 0 to 10 with 0 being the lowest level of pain and 10 being the highest level of pain . The patient identifies his level of pain on this graduated line.
Evaluation of Analgesic effect of at least 30% | 12 months
  Percentage of patients with at least 30% of pain reduction base on numeric scale within the last week before the end of treatment. Pain intensity will be measured using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of pain and 10 being the highest level of pain. The patient identifies his level of pain on this graduated line.
Evaluation of Severe Adverse Events (SAE) | over the 12 months
  Declaration of all severe adverse event occurring during the 12 months period of treatment. Each event will be analyzed by an independent committee to evaluate the immutability of the experimental treatment.
Evaluation of patient satisfaction with pain treatment at first visit to refill the pump (1 month) assessed by the Visual Analogic Scale (VAS) | 1 month
  Satisfaction level of patient's pain relief will be assessed using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of satisfaction and 10 being the highest satisfaction. The patient identifies his level of satisfaction of pain relief on this graduated line.
Evaluation patient satisfaction of pain relief with the treatment at 6 months assessed by the Visual Analogic Scale (VAS) | 6 months
  Satisfaction level of patient's pain relief will be assessed using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of satisfaction and 10 being the highest satisfaction. The patient identifies his level of satisfaction of pain relief on this graduated line.
Evaluation patient satisfaction of pain relief with the treatment 12 months assessed by the Visual Analogic Scale (VAS) | 12 months
  Satisfaction level of patient's pain relief will be assessed using visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of satisfaction and 10 being the highest satisfaction. The patient identifies his level of satisfaction of pain relief on this graduated line.
Analgesic effect on spontaneous pain duration | 1 month before initiation of treatment
  Duration (average time per day)
Analgesic effect on spontaneous pain duration | 6 months
  Duration (average time per day)
Analgesic effect on spontaneous pain duration | 12 months
  Duration (average time per day)
Analgesic effect on spontaneous pain intensity | 1 month before initiation of treatment
  Intensity of spontaneous pain will be assessed using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of intensity of pain and 10 being the highest intensity of pain. The patient identifies his level of pain intensity on this graduated line.
Analgesic effect on spontaneous pain intensity | initial evaluation 6 months
  intensity (numeric scale) of spontaneous pain. This numeric scale is a graduated line from 0 to 10, 0 being the lowest level of intensity of pain and 10 being the highest intensity of pain. T The patient identifies his level of pain intensity on this graduated line.
Analgesic effect on spontaneous pain intensity | initial evaluation 12 months
  intensity (numeric scale) of spontaneous pain. This numeric scale is a graduated line from 0 to 10, 0 being the lowest level of pain intensity and 10 being the highest pain intensity. The patient identifies his level of pain intensity on this graduated line.
Analgesic effect on provoked pain duration | initial evaluation
  Duration (average time per day)
Analgesic effect on provoked pain duration | 6 months
  Duration (average time per day)
Analgesic effect on provoked pain duration | 12 months
  Duration (average time per day)
Analgesic effect on provoked pain intensity | 1 month before initiation of treatment
  Intensity of provoked pain will be assessed using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of pain intensity and 10 being the highest pain intensity.
Analgesic effect on provoked pain intensity | 6 months
  intensity of provoked pain will be assessed using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of pain intensity and 10 being the highest pain intensity.
Analgesic effect on provoked pain intensity | 12 months
  intensity of provoked pain will be assessed using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of pain intensity and 10 being the highest pain intensity.
Quality of life at inclusion assessed by the Short Form questionnaire (SF12) | 1 month before initiation of treatment
  Quality of life will be assessed using the 12 items Short Form questionnaire (SF12). It is a self-reported multipurpose questionnaire generic measure of health status. It measure in 12 questions, 8 concepts: physical functioning, role limitation due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. A specific algorithm gives a standardized total score between 0 and 100 for physical and mental summary scale. The higher the score, the better the quality of life.
Quality of life at 6 months assessed by the Short Form questionnaire (SF12) | 6 months
  Quality of life will be assessed using the 12 items Short Form questionnaire (SF12). It is a self-reported multipurpose questionnaire generic measure of health status. It measure in 12 questions, 8 concepts: physical functioning, role limitation due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. A specific algorithm gives a standardized total score between 0 and 100 for physical and mental summary scale. The higher the score, the better the quality of life.
Quality of life at 12 months assessed by the Short Form questionnaire (SF12) | 12 months
  Quality of life will be assessed using the 12 items Short Form questionnaire (SF12). It is a self-reported multipurpose questionnaire generic measure of health status. It measure in 12 questions, 8 concepts: physical functioning, role limitation due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. A specific algorithm gives a standardized total score between 0 and 100 for physical and mental summary scale. The higher the score, the better the quality of life.
Patient global impression of change | at one months of treatment (first refill of the pump)
  Patient global impression of change estimated using a using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of pain intensity and 10 being the highest pain intensity.
Patient global impression of change | 6 months
  Patient global impression of change estimated using a using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of pain intensity and 10 being the highest pain intensity.
Patient global impression of change | 12 months
  Patient global impression of change estimated using a visual analogic scale (VAS). This VAS is a graduated line from 0 to 10, 0 being the lowest level of pain intensity and 10 being the highest pain intensity.
Analgesic drugs intake at inclusion | 1 month before initiation of treatment
  Quantification of analgesic drugs intake per day with differentiation of class of analgesics.
Analgesic drugs intake at 12 months | 12 months
  Quantification of analgesic drugs intake per day with differentiation of class of analgesics.
Evaluation of cognition effects induced by ITZ at inclusion | 1 month before initiation of treatment
  Mini Mental State Examination (MMSE) questionnaire will be used to evaluate cognition effect. Each 30 questions is one point. Patients with score greater than 27 has no mental issue, between 24 et 27 light dementia, less than 24 dementia.
Evaluation of cognition effects induced by ITZ at 6 months | 6 months
  Mini Mental State Examination (MMSE) questionnaire will be used to evaluate cognition effect. Each 30 questions is one point. Patients with score greater than 27 has no mental issue, between 24 et 27 light dementia, less than 24 dementia.
Evaluation of cognition effects induced by ITZ at 12 months | 12 months
  Mini Mental State Examination (MMSE) questionnaire will be used to evaluate cognition effect. Each 30 questions is one point. Patients with score greater than 27 has no mental issue, between 24 et 27 light dementia, less than 24 dementia.
Measure of neuro- psychological effects of depression induced by ITZ | 1 month before initiation of treatment
  Hospital Anxiety and Depression Scale (HADS) for depression include 7 questions with a score from 0 to 3. If the score is greater than 11 then the patient suffer from depression
Measure of neuro- psychological effects of depression induced by ITZ | 6 months
  Hospital Anxiety and Depression Scale (HADS) for depression include 7 questions with a score from 0 to 3. If the score is greater than 11 then the patient suffer from depression
Measure of neuro- psychological effects of depression induced by ITZ | 12 months
  Hospital Anxiety and Depression Scale (HADS) for depression include 7 questions with a score from 0 to 3. If the score is greater than 11 then the patient suffer from depression
Measure of neuro- psychological anxiety effects induced by ITZ | 1 month before initiation of treatment
  Hospital Anxiety and Depression Scale (HADS) for anxiety include 7 questions with a score from 0 to 3. If the score is greater than 11 then the patient suffer from anxiety.
Measure of neuro- psychological anxiety effects induced by ITZ | 6 months
  Hospital Anxiety and Depression Scale (HADS) for anxiety include 7 questions with a score from 0 to 3. If the score is greater than 11 then the patient suffer from anxiety.
Measure of neuro- psychological anxiety effects induced by ITZ | 12 months
  Hospital Anxiety and Depression Scale (HADS) for anxiety include 7 questions with a score from 0 to 3. If the score is greater than 11 then the patient suffer from anxiety.
Impact of ITZ on psycho-social status of patients | 1 month before initiation of treatment
  Pain catastrophizing scale (PCS) score to assess the patient's physical and emotional distress associated with their pain condition. The scale is composed of 13 questions with a score for each questions going from 0 to 4. The final score is the addition of the score of each question, going from 0 to 52. Patient with a score greater than the 75% percentile mean value is at high risk of pain chronicity. Patient with a score between the 50 % and 75% percentile mean value is at moderate risk of pain chronicity
Impact of ITZ on psycho-social status of patients | 6 months
  Pain catastrophizing scale (PCS) score to assess the patient's physical and emotional distress associated with their pain condition. The scale is composed of 13 questions with a score for each questions going from 0 to 4. The final score is the addition of the score of each question, going from 0 to 52. Patient with a score greater than the 75% percentile mean value is at high risk of pain chronicity. Patient with a score between the 50 % and 75% percentile mean value is at moderate risk of pain chronicity
Impact of ITZ on psycho-social status of patients | 12 months
  Pain catastrophizing scale (PCS) score to assess the patient's physical and emotional distress associated with their pain condition. The scale is composed of 13 questions with a score for each questions going from 0 to 4. The final score is the addition of the score of each question, going from 0 to 52. Patient with a score greater than the 75% percentile mean value is at high risk of pain chronicity. Patient with a score between the 50 % and 75% percentile mean value is at moderate risk of pain chronicity

CONTACTS AND LOCATIONS:
Overall Officials: MERTENS Patrick, MD, PhD, Study Director — Hospices Civils de Lyon

IPD SHARING:
Plan to Share IPD: No